CLINICAL TRIAL: NCT05696704
Title: Utilizing Telehealth to Reduce Pre-Death Grief, Burden, and Stress in Family Caregivers
Brief Title: Telehealth to Reduce Mental Health in Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TexasTechU2
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Issue; Grief; Burden, Caregiver
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy (MBCT) combines the ideas of cognitive therapy with meditative practices and attitudes based on the cultivation of mindfulness. The heart of this work lies in becoming acquainted with the modes of mind that often characterize mood disorders while simultaneously learning to develop a new relationship to them.
  Interventions: Other: Behavioral: Mindfulness Based Cognitive Therapy
- Behavior Activation (Experimental): BA Increase reinforcing behaviors in order to influence emotions and cognitions.
  Interventions: Other: Behavioral: Behavior Activation

INTERVENTIONS:
Other: Behavioral: Mindfulness Based Cognitive Therapy — Individual tele-therapy 12 to 16 weeks
  Other Names: MBCT
  Arms: Mindfulness Based Cognitive Therapy
Other: Behavioral: Behavior Activation — Individual therapy 12 to 16 weeks
  Other Names: BA
  Arms: Behavior Activation

SUMMARY:
The overarching goal of this project is to evaluate if evidence-based interventions can reduce PDG, burden, and stress in informal caregivers of individuals with dementia when provided over telehealth.

DETAILED DESCRIPTION:
Aim 1: Examine the effects of two individual evidence-based therapies for informal caregivers of dementia patients over telehealth.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be informal caregivers (e.g., spouse; child; close friend) of individuals with dementia
* Informal caregivers can be family members or close friends
* Adults (18 to 89 years old) who read, write, and speak in English
* Mental Health Diagnosis (e.g., Generalized Anxiety Disorder; Major Depressive Disorder

Exclusion Criteria:

* Formal caregivers (who are being paid to take care of the patient)
* Any informal caregivers with cognitive impairment is identified during the assessment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief Scale-12 (measuring pre-death grief) | [Time Frame: through study completion, an average of 6 months]
  The PG-12 (range 11-55; higher scores mean higher pre-death grief), which is used to measure pre-death grief will be used to measure grief of having a loved one live with a life limiting illness and no longer be able to engage in valued activities.

SECONDARY OUTCOMES:
Zarit Burden Inventory (ZBI) | [Time Frame: through study completion, an average of 6 months]
  Informal caregivers, usually family member, have an increase in burden or feeling they are overwhelmed by their current circumstances. The ZBI is between 0-48, higher scores indicating higher burden.
Perceived Stress Scale | [Time Frame: through study completion, an average of 6 months]
  Informal caregivers, usually family members, are unpaid and have a tendency to feel tense and emotionally drained do to caregiving. Scores range from 0-40 with higher scores indicating higher rates of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Singer, Ph.D., Principal Investigator — jonsinge@ttu.edu
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No